CLINICAL TRIAL: NCT01633164
Title: Re-Inventing Yourself After SCI: A Site-Specific Randomized Clinical Trial
Brief Title: Re-Inventing Yourself After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H133N110006
Record Dates: First submitted 2012-06-26; First posted 2012-07-04 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Self-Efficacy; Life Satisfaction; Community Participation
MeSH Terms: conditions — Spinal Cord Injuries; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCI Reinvention Protocol Participants (Experimental): This group will receive 6 instructor-led 2 hour long didactic presentations regarding 8 key principles of self-efficacy and experiential exercises, including goal setting and problem solving with extensive group discussion. At the end of each session, tasks are assigned to participants to be completed outside the group during the week between sessions. Experiences from these activities and practice implementing the intervention principles will be shared and discussed each week, providing additional opportunities for problem solving and positive feedback.
  Interventions: Behavioral: SCI Reinvention Protocol Participants
- Waitlist Group (Other): This group will include individuals randomized to receive no treatment for the 30 weeks during which the interventional group will receive the active treatment and have their progress tracked.
  Interventions: Other: Waitlist Group

INTERVENTIONS:
Behavioral: SCI Reinvention Protocol Participants — The intervention involves participation in a six week psychologically-based educational intervention. During the course, 8 specific skills are reviewed in order to specifically address reframing a person's method of looking at events, build confidence by focusing on personal strengths, develop methods of recognizing and appreciating the good in one's life and express gratitude for positive attributes. These skills are presented in a specific sequence so that participants can gain mastery of introductory concepts before undertaking those that are both more difficult and complex.
  Arms: SCI Reinvention Protocol Participants
Other: Waitlist Group — Wait list arm will begin study intervention after 4 1/2 months.
  Arms: Waitlist Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of a replicable, psychologically-based group education intervention, Re-Inventing Yourself after Spinal Cord Injury (SCI), which aims to enhance personal self-efficacy. A structured six-week, manualized, group therapy intervention that delivers positive psychology concepts within a cognitive-behavioral therapy-based model has been created for the purpose of developing a resilient and optimistic sense of efficacy for people with SCI. Concepts covered within this intervention include: reframing and restructuring a person's method of looking at events, building confidence by focusing on personal strengths, developing methods of recognizing and appreciating the good in one's life and expressing gratitude for positive attributes. The goals of this intervention are to increase personal self-efficacy, enhance emotional well-being and improve participation in society for people with SCI living in the community. The investigators hypothesize that persons receiving the intervention will demonstrate improved SCI-specific and overall self-efficacy as compared to waitlist controls.

ELIGIBILITY:
Inclusion Criteria:

1. History of traumatic SCI at any level;
2. at least 4 weeks post-discharge from initial inpatient rehabilitation;
3. 18 years of age or older at the time of study enrollment;
4. English speaking in order to complete study measures and participate in group interactions; and
5. able to provide informed consent to participate

Exclusion Criteria:

1. History of moderate or severe traumatic brain injury;
2. current participation in another RCT;
3. live beyond a reasonable commuting distance from Craig Hospital;
4. unable to verbally communicate;
5. unable to attend group sessions;
6. active participation in another formal clinical group or psychological therapy;
7. are currently experiencing moderately severe or greater levels of depression which would require more intense treatment than is provided in this intervention, as evidenced by a score of 15 or higher on the Personal Health Questionnaire-9;37
8. are currently of high self efficacy, as determined by a score of 90 or higher on the MSES,32 which has a range of 16 to 112, with higher scores representing higher SCI-specific self-efficacy; or
9. have any condition that, in the judgment of the investigators, precludes successful participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Moorong Self-Efficacy Scale (MSES) score over a 30 week time period | Baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  The MSES is a 16 item self-report measure of self-efficacy related to everyday life activities, designed specifically for persons with SCI. Individuals use a 7-point Likert scale ranging from 1 (very uncertain) to 7 (very certain) to rate their ability to perform 16 everyday tasks, with higher scores representing greater perceived self-efficacy.

SECONDARY OUTCOMES:
Change in General Self-Efficacy Scale scores over a 30 week time period | Baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  The General Self-Efficacy Scale (GSES) is a questionnaire designed to assess a person's ability to cope with a variety of difficult demands in life, with ten items scored using a Likert rating scale, ranging from 1 (not at all true) to 4 (exactly true).

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States